CLINICAL TRIAL: NCT01905748
Title: Acute Phase Reactions and Thrombophilia in Pediatric Patients With Migraine, Laboratory Investigations in Steady State and During Migraine Attack
Brief Title: Acute Phase Reactions and Thrombophilia in Pediatric Patients With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dpt B and Pediatric Hematology Unit, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0040-09-EMC
Record Dates: First submitted 2011-09-27; First posted 2013-07-23 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Migraine; Thrombophilia
Keywords: Coagulation
MeSH Terms: conditions — Migraine Disorders; Thrombophilia; Thrombosis | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients during Migraine attacks (Experimental): Patients with Migraine before, during and after Migraine attacks. Acute phase reaction profile, and activation of the coagulation system will be investigated together with thrombophilia profile.
  Interventions: Other: Laboratory tests
- Control group (Experimental): Patients with acute neurologic events like convulsions not related to fever or central nervous system (CNS) infections will be studied including acute phase reaction laboratory tests, thrombophilia and activation of the coagulation system
  Interventions: Other: Laboratory tests

INTERVENTIONS:
Other: Laboratory tests — Laboratory tests: erythrocyte sedimentation rate (ESR), Blood Count, C reactive Protein, Protein C activity, Protein S activity,Antithrombin II activity, Coagulation Factor VIII and IX,Con Willebrand Factor, prothrombin time (PT), activated partial thromboplastin time (aPTT), Fibrinogen, D Dimer and Prothrombin Fragments F1 and F2.

SUMMARY:
Acute Migraine attacks can be related to vascular or coagulation activation. Previous studies found relative high incidence of prothrombotic events in Migraine. The present study intends to assess the coagulation system and activation in patients with Migraine during steady state phase and at the beginning of attacks and after 72 hours. A control group of patients with another acute neurologic event like convulsions will be also studied. Patients will be at pediatric age and teenagers.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the pediatric age (5 to 20 ys old) suffering from Migraine attacks diagnosed by a neurologist.

Exclusion Criteria:

* Patients with other underlying neurological conditions of coagulation diseases

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-08; Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with activation of the coagulation system. | Two years, each patient will be studied at attack onset and after 72 hours.
  The further analysis will be performed in each patient: Pt, PTT, Platelets, Protein C, S, Antithrombin III, D Dimer, Factor VIII, Factor IX, Von Willebrand Factor and Prothrombin fragments I and II will be analyzed on day one of the crises, after 72 hours and in steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Ha'Emek Medical Center, Afula, Israel